CLINICAL TRIAL: NCT05363163
Title: Clinical Study for the Effectiveness of Use of an Injectable Medical Device GANA X® in the Treatment of Buttocks Volume Depression
Brief Title: Clinical Study for the Evaluation of the Effectiveness of Use of a Poly-L Lactic Acid Injectable Filler for the Aesthetic Treatment of Buttocks Volume Depression
Acronym: PLLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Co., Ltd (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E0805; 2021-A02728-33 (Other: ANSM)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Buttocks Volume Loss

STUDY DESIGN:
Intervention Model Description: All participants will receive the same medical device (Gana X)
Masking Description: Participants and investigators assessors will know which filler was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gana X (Experimental): Participants will receive Gana X in both buttocks
  Interventions: Device: Gana X

INTERVENTIONS:
Device: Gana X — Injection in the deep dermis and subcutaneous layer of the buttocks on D0 (initial injection) and 1 month and a half after initial injection if necessary (optional touch-up).

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of Gana X, a Poly L-lactic acid filler for the aesthetic treatment of buttocks.

DETAILED DESCRIPTION:
A screening visit will allow to inform and preselect the participants.

On D0, baseline scoring, fringe projection acquisitions and photographs will be done before injection. Eligible participants will receive a first injection of the product. Immediately after injection, injector's treatment satisfaction will be collected. Investigator evaluator will collect Adverse Events (AEs) and Injection Site Reactions (ISRs) immediately after injection.

A month and a half after initial injection (M1 and a half), clinical scoring, fringe projection acquisitions and photographs will be done before touch-up (if applicable). Participant's treatment satisfaction and injector's treatment satisfaction (if applicable) will be collected. A touch-up injection will be made if necessary, according to injector and participant opinion. Investigator evaluator will collect AEs and ISRs before and after touch-up if applicable.

Six (M6), nine (M9), twelve (M12), eighteen (M18) and twenty-four (M24) months after initial injection, clinical scoring, fringe projection acquisitions and photographs will be done. Participant's treatment satisfaction will be collected. Investigator evaluator will collect AEs and ISRs.

ELIGIBILITY:
Inclusion Criteria:

* Subject with mild to moderate buttock volume depression and/or seeking buttocks volume augmentation based on investigator evaluation.
* Subject wiling to abstain from other body contouring procedures during the whole study period.
* Subject psychologically able to understand the study related information and to give a written informed consent.
* Subject having given freely and expressly his/her informed consent.
* Subject willing to have photographs taken.
* Subject affiliated to a health social security system.
* Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit and during the whole study period.

Exclusion Criteria:

* Pregnant or nursing woman or having given birth within the last year or planning a pregnancy during the study.
* Excessive subcutaneous fat in the area to be treated.
* Excessive skin laxity on the area to be treated.
* Severe buttocks ptosis.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment
* Subject participation to another research on human beings or who is in an exclusion period of one.
* Subject having already received 4500 euros indemnities for participation in research involving human beings in the 12 previous months or exceeding these 4500 euros with his participation in the present study.
* Subject suspected to be non-compliant according to the investigator's judgment.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject with a history of cellulitis, streptococcal disease, such as acute rheumatic fever or recurrent sore throats and in case of acute rheumatic fever with heart complications.
* Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (e.g. acne, chronic eczema, atopic dermatitis…).
* Subject with an abscess, unhealed wound, or a cancerous or precancerous lesion on the studied zone.
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Subject with a tendency to develop keloids or hypertrophic scarring.
* Subject with significant scarring, open wounds, lesions or tattoos in or near the area to be treated.
* Subject having history of allergy or anaphylactic shock including hypersensitivity to Poly-l-lactic acid, to lidocaine or to one of the components of the tested devices or antiseptic solution.
* Subject having received a dose of COVID-19 vaccine within the 14 days prior to injection visits or planning to receive a dose in the 14 days following injections.
* Subject having received treatment on or near the buttocks (laser, dermabrasion, surgery, radiofrequency, cryolipolysis, buttocks electrostimulation, endermologie, liposuction, other energy-based treatment, surgery…) within the 12 months prior to screening visit.
* Subject having received injection with a resorbable filling product in or near the buttocks within the 12 months prior to screening visit.
* Subject having received at any time the following treatments in the area to be treated:

  * Buttocks implants;
  * Buttocks fillers (e.g., silicone, semi-permanent or permanent fillers or autologous fat injections);
  * Injections for the treatment of cellulitis.
* Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.
* Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAID) (ibuprofen, naproxen, …), antiplatelet agents, anticoagulants or other substances known to prolong bleeding time within 1 week prior to injection visits.
* Subject undergoing a topical treatment on the test area or a systemic treatment:

  * Antihistamines during the 2 weeks prior to injections visits (D0 and touch-up visit).
  * Immunosuppressors and/or corticoids during the 4 weeks prior to injections visits (D0 and touch-up visit).
  * Retinoids during the 6 months prior to injections visits (D0 and touch-up visit).
* Intensive exposure to sunlight or UV-rays within the month before injection visits and one month after.
* Subject planning to loss or gain weight for the duration of the study.
* Subject planning to change her/his life habits during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation was initiated on 2 May 2022 (first subject first visit). Subjects were recruited from one investigational center, in France. The last subject was screened on 7 November 2022 and the recruitment period lasted 189 days.
Pre-assignment Details: 126 subjects were screened to randomize 50 subjects
Groups:
- Gana X: Participants received Gana X in both buttocks using injection in the deep dermis and subcutaneous layer of the buttocks on D0 (initial injection) and 1 month and a half after initial injection if necessary (optional touch-up).
Period: Overall Study
Arm/Group | Gana X
Started | 50
Completed | 37
Not Completed | 13
Not completed — Withdrawal by Subject | 13

BASELINE CHARACTERISTICS:
Groups:
- Gana X: Participants received Gana X in both buttocks
Arm/Group | Gana X
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.06 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Buttocks Volume 6 Months After Treatment
Description: This will be assessed using 3D acquisitions of the buttocks analysed on a computer software to evaluate the decrease of the buttocks hollow. To observe an improvement, an increase of the mean change from baseline value was expected.
Time Frame: Baseline and Month 6
Population: Intent To Treat population - any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Gana X
Number analyzed (Participants) | 47
cm^3 | 22.21 (11.65)
Statistical Analysis 1: Comparison: Gana X; Test type: Other — If the mean volume variation was higher than 0 and the p-value of the statistical test lower than 0.05, the H0 hypothesis was rejected, and the primary endpoint demonstrated; p < 0.0001, t-test, 2 sided — p-value of the statistical test lower than 0.05

2. Secondary Outcome: Change From Baseline in Buttocks Volume
Description: as for outcome 1
Time Frame: Baseline, Month 1^1/2, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Gana X
Number analyzed (Participants) | 50
cm^3
  Change from baseline (D0 visit) to M11/2 visit | 11.99 (7.73)
  Change from baseline (D0 visit) to M9 visit: number analyzed (Participants) | 40
  Change from baseline (D0 visit) to M9 visit | 21.70 (12.14)
  Change from baseline (D0 visit) to M12 visit: number analyzed (Participants) | 39
  Change from baseline (D0 visit) to M12 visit | 22.29 (13.38)
  Change from baseline (D0 visit) to M18 visit: number analyzed (Participants) | 36
  Change from baseline (D0 visit) to M18 visit | 16.95 (11.60)
  Change from baseline (D0 visit) to M24 visit: number analyzed (Participants) | 36
  Change from baseline (D0 visit) to M24 visit | 10.96 (10.21)

3. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Responder Rate
Description: Percentage of participants with an improvement on GAIS. A responder is defined as a subject having "Improved", "Much improved" or "Very much improved" score according to GAIS.
Time Frame: Month 1^1/2, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included in the study with at least a post-basal value.
Measure: Count of Participants; unit: Participants
Arm/Group | Gana X
Number analyzed (Participants) | 50
Participants
  Evaluated by the independent blind evaluator at M11/2: Responder | 36
  Evaluated by the independent blind evaluator at M11/2: Not Responder | 14
  Evaluated by the independent blind evaluator at M6: number analyzed (Participants) | 47
  Evaluated by the independent blind evaluator at M6: Responder | 46
  Evaluated by the independent blind evaluator at M6: Not Responder | 1
  Evaluated by the independent blind evaluator at M9: number analyzed (Participants) | 40
  Evaluated by the independent blind evaluator at M9: Responder | 38
  Evaluated by the independent blind evaluator at M9: Not Responder | 2
  Evaluated by the independent blind evaluator at M12: number analyzed (Participants) | 39
  Evaluated by the independent blind evaluator at M12: Responder | 37
  Evaluated by the independent blind evaluator at M12: Not Responder | 2
  Evaluated by the independent blind evaluator at M18: number analyzed (Participants) | 35
  Evaluated by the independent blind evaluator at M18: Responder | 26
  Evaluated by the independent blind evaluator at M18: Not Responder | 9
  Evaluated by the independent blind evaluator at M24: number analyzed (Participants) | 37
  Evaluated by the independent blind evaluator at M24: Responder | 26
  Evaluated by the independent blind evaluator at M24: Not Responder | 11
  Evaluated by the subject at M11/2: number analyzed (Participants) | 49
  Evaluated by the subject at M11/2: Responder | 27
  Evaluated by the subject at M11/2: Not Responder | 22
  Evaluated by the subject at M6: number analyzed (Participants) | 47
  Evaluated by the subject at M6: Responder | 42
  Evaluated by the subject at M6: Not Responder | 5
  Evaluated by the subject at M9: number analyzed (Participants) | 38
  Evaluated by the subject at M9: Responder | 32
  Evaluated by the subject at M9: Not Responder | 6
  Evaluated by the subject at M12: number analyzed (Participants) | 38
  Evaluated by the subject at M12: Responder | 33
  Evaluated by the subject at M12: Not Responder | 5
  Evaluated by the subject at M18: number analyzed (Participants) | 36
  Evaluated by the subject at M18: Responder | 29
  Evaluated by the subject at M18: Not Responder | 7
  Evaluated by the subject at M24: number analyzed (Participants) | 37
  Evaluated by the subject at M24: Responder | 28
  Evaluated by the subject at M24: Not Responder | 9

4. Secondary Outcome: Percentage of Satisfied Participants
Description: Percentage of participants with positive answers to an internal questionnaire
Time Frame: Month 1^1/2, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included in the study with at least a post-basal value
Measure: Count of Participants; unit: Participants
Arm/Group | Gana X
Number analyzed (Participants) | 50
Participants
  Are you satisfied with how your buttocks looks at M11/2?: Satisfied | 31
  Are you satisfied with how your buttocks looks at M11/2?: Not satisfied | 19
  Are you satisfied with how your buttocks looks at M6?: number analyzed (Participants) | 47
  Are you satisfied with how your buttocks looks at M6?: Satisfied | 39
  Are you satisfied with how your buttocks looks at M6?: Not satisfied | 8
  Are you satisfied with how your buttocks looks at M9?: number analyzed (Participants) | 40
  Are you satisfied with how your buttocks looks at M9?: Satisfied | 33
  Are you satisfied with how your buttocks looks at M9?: Not satisfied | 7
  Are you satisfied with how your buttocks looks at M12?: number analyzed (Participants) | 39
  Are you satisfied with how your buttocks looks at M12?: Satisfied | 33
  Are you satisfied with how your buttocks looks at M12?: Not satisfied | 6
  Are you satisfied with how your buttocks looks at M18?: number analyzed (Participants) | 36
  Are you satisfied with how your buttocks looks at M18?: Satisfied | 31
  Are you satisfied with how your buttocks looks at M18?: Not satisfied | 5
  Are you satisfied with how your buttocks looks at M24?: number analyzed (Participants) | 37
  Are you satisfied with how your buttocks looks at M24?: Satisfied | 32
  Are you satisfied with how your buttocks looks at M24?: Not satisfied | 5
  The result is aesthetically satisfying at M11/2: Satisfied | 33
  The result is aesthetically satisfying at M11/2: Not satisfied | 17
  The result is aesthetically satisfying at M6: number analyzed (Participants) | 47
  The result is aesthetically satisfying at M6: Satisfied | 40
  The result is aesthetically satisfying at M6: Not satisfied | 7
  The result is aesthetically satisfying at M9: number analyzed (Participants) | 40
  The result is aesthetically satisfying at M9: Satisfied | 32
  The result is aesthetically satisfying at M9: Not satisfied | 8
  The result is aesthetically satisfying at M12: number analyzed (Participants) | 38
  The result is aesthetically satisfying at M12: Satisfied | 32
  The result is aesthetically satisfying at M12: Not satisfied | 6
  The result is aesthetically satisfying at M18: number analyzed (Participants) | 36
  The result is aesthetically satisfying at M18: Satisfied | 30
  The result is aesthetically satisfying at M18: Not satisfied | 6
  The result is aesthetically satisfying at M24: number analyzed (Participants) | 37
  The result is aesthetically satisfying at M24: Satisfied | 32
  The result is aesthetically satisfying at M24: Not satisfied | 5
  The result is natural at M11/2: Satisfied | 41
  The result is natural at M11/2: Not satisfied | 9
  The result is natural at M6: number analyzed (Participants) | 47
  The result is natural at M6: Satisfied | 44
  The result is natural at M6: Not satisfied | 3
  The result is natural at M9: number analyzed (Participants) | 40
  The result is natural at M9: Satisfied | 37
  The result is natural at M9: Not satisfied | 3
  The result is natural at M12: number analyzed (Participants) | 38
  The result is natural at M12: Satisfied | 31
  The result is natural at M12: Not satisfied | 7
  The result is natural at M18: number analyzed (Participants) | 36
  The result is natural at M18: Satisfied | 35
  The result is natural at M18: Not satisfied | 1
  The result is natural at M24: number analyzed (Participants) | 37
  The result is natural at M24: Satisfied | 35
  The result is natural at M24: Not satisfied | 2
  The buttocks volume are restored at M11/2: number analyzed (Participants) | 49
  The buttocks volume are restored at M11/2: Satisfied | 31
  The buttocks volume are restored at M11/2: Not satisfied | 18
  The buttocks volume are restored at M6: number analyzed (Participants) | 47
  The buttocks volume are restored at M6: Satisfied | 39
  The buttocks volume are restored at M6: Not satisfied | 8
  The buttocks volume are restored at M9: number analyzed (Participants) | 40
  The buttocks volume are restored at M9: Satisfied | 30
  The buttocks volume are restored at M9: Not satisfied | 10
  The buttocks volume are restored at M12: number analyzed (Participants) | 38
  The buttocks volume are restored at M12: Satisfied | 31
  The buttocks volume are restored at M12: Not satisfied | 7
  The buttocks volume are restored at M18: number analyzed (Participants) | 36
  The buttocks volume are restored at M18: Satisfied | 28
  The buttocks volume are restored at M18: Not satisfied | 8
  The buttocks volume are restored at M24: number analyzed (Participants) | 37
  The buttocks volume are restored at M24: Satisfied | 29
  The buttocks volume are restored at M24: Not satisfied | 8
  The buttocks skin laxity is improved at M11/2: Satisfied | 30
  The buttocks skin laxity is improved at M11/2: Not satisfied | 20
  The buttocks skin laxity is improved at M6: number analyzed (Participants) | 47
  The buttocks skin laxity is improved at M6: Satisfied | 33
  The buttocks skin laxity is improved at M6: Not satisfied | 14
  The buttocks skin laxity is improved at M9: number analyzed (Participants) | 40
  The buttocks skin laxity is improved at M9: Satisfied | 29
  The buttocks skin laxity is improved at M9: Not satisfied | 11
  The buttocks skin laxity is improved at M12: number analyzed (Participants) | 38
  The buttocks skin laxity is improved at M12: Satisfied | 31
  The buttocks skin laxity is improved at M12: Not satisfied | 7
  The buttocks skin laxity is improved at M18: number analyzed (Participants) | 36
  The buttocks skin laxity is improved at M18: Satisfied | 27
  The buttocks skin laxity is improved at M18: Not satisfied | 9
  The buttocks skin laxity is improved at M24: number analyzed (Participants) | 37
  The buttocks skin laxity is improved at M24: Satisfied | 30
  The buttocks skin laxity is improved at M24: Not satisfied | 7

5. Secondary Outcome: Injector Satisfaction
Description: The investigator who will inject the product will complete a questionnaire for each participant.
Time Frame: After initial injection (Day 0)
Population: Intent To Treat population - any subject included in the study with at least a post-basal value
Measure: Count of Participants; unit: Participants
Arm/Group | Gana X
Number analyzed (Participants) | 50
Participants
  Ease of injection: Very satisfied | 34
  Ease of injection: satisfied | 13
  Ease of injection: Somewhat satisfied | 2
  Ease of injection: Somewhat dissatisfied | 1
  Ease of injection: Dissatisfied | 0
  Ease of injection: Very dissatisfied | 0
  Mouldability: Very satisfied | 28
  Mouldability: satisfied | 21
  Mouldability: Somewhat satisfied | 1
  Mouldability: Somewhat dissatisfied | 0
  Mouldability: Dissatisfied | 0
  Mouldability: Very dissatisfied | 0
  Ease of product positioning: Very satisfied | 29
  Ease of product positioning: satisfied | 14
  Ease of product positioning: Somewhat satisfied | 7
  Ease of product positioning: Somewhat dissatisfied | 0
  Ease of product positioning: Dissatisfied | 0
  Ease of product positioning: Very dissatisfied | 0
  Immediate result: Very satisfied | 22
  Immediate result: satisfied | 18
  Immediate result: Somewhat satisfied | 9
  Immediate result: Somewhat dissatisfied | 1
  Immediate result: Dissatisfied | 0
  Immediate result: Very dissatisfied | 0
  Result after massage: Very satisfied | 23
  Result after massage: satisfied | 23
  Result after massage: Somewhat satisfied | 4
  Result after massage: Somewhat dissatisfied | 0
  Result after massage: Dissatisfied | 0
  Result after massage: Very dissatisfied | 0

6. Secondary Outcome: Collection of Injection Site Reactions
Description: Injection site reactions are usual signs reported after injection and consist on the evaluation of the following signs : Redness / Erythema, Pain / Tenderness, Induration / Firmness, Swelling / Edema, Lumps / Bumps, Bruising, Itching, Coloration, Pigmentation / Discoloration.
  Data presented are a percentage of subjects presenting at least one ISR of any severity evaluated by the investigator
Time Frame: Day 0, Month 1^1/2, Month 6, Month 9, Month 12, Month 18 and Month 24]
Population: Safety population - any subject having used the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Gana X
Number analyzed (Participants) | 50
Participants
  D0 after initial injection: At least one sign | 32
  D0 after initial injection: No sign | 18
  M11/2 before touch-up: At least one sign | 2
  M11/2 before touch-up: No sign | 48
  M11/2 after touch-up: number analyzed (Participants) | 45
  M11/2 after touch-up: At least one sign | 40
  M11/2 after touch-up: No sign | 5
  M6: number analyzed (Participants) | 47
  M6: At least one sign | 7
  M6: No sign | 40
  M9: number analyzed (Participants) | 40
  M9: At least one sign | 4
  M9: No sign | 36
  M12: number analyzed (Participants) | 39
  M12: At least one sign | 6
  M12: No sign | 33
  M18: number analyzed (Participants) | 36
  M18: At least one sign | 9
  M18: No sign | 27
  M24: number analyzed (Participants) | 37
  M24: At least one sign | 6
  M24: No sign | 31

7. Secondary Outcome: Collection of Adverse Events
Description: Number of Adverse Events (AEs) Number of Adverse Device Effects (ADEs) Percentage of subjects with at least one AE Percentage of subject with at least one ADE
Time Frame: Day 0 to Month 24
Population: Safety population - any subject having used the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Gana X
Number analyzed (Participants) | 50
Participants
  Subjects with at least one AE:: With | 39
  Subjects with at least one AE:: Without | 11
  Subjects with at least one SAE:: With | 1
  Subjects with at least one SAE:: Without | 49
  subjects with at least one ADE:: With | 28
  subjects with at least one ADE:: Without | 22
  Subjects with at least one SADE:: With | 0
  Subjects with at least one SADE:: Without | 50

ADVERSE EVENTS:
Time Frame: 24 months
Description: Definitions from MDCG were used as the study was done on a medical device
Arm/Group | Gana X
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gana X (N=50)
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gana X (N=50)
Headache (Nervous system disorders) | 18 (67)
Angina (Infections and infestations) | 3 (3)
Dysmenorrhea (General disorders) | 4 (15)
Lump/nodule (Product Issues) | 8 (9)
Pain (General disorders) | 17 (25)

LIMITATIONS AND CAVEATS:
The number of injections sessions was quite low in this clinical investigation and is thus not representative of the usual medical practice. However, in most of the publications presenting efficacy and safety of PLLA in Buttocks, 1 to 3 sessions were done

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05363163/Prot_SAP_000.pdf